CLINICAL TRIAL: NCT06235502
Title: A Cluster Randomised Controlled Trial on the Effects of Long-term Home-based Exercise for Patients With Chronic Obstructive Pulmonary Disease With Recent Exacerbation: the COPDtoParis Project
Brief Title: Long-term Home-based Exercise for Patients With COPD: the COPDtoParis Project
Acronym: COPDtoParis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Karen Elise Jensen Foundation (Other); Simon Fougners Hartmann Family Foundation (Unknown); 4Mvideo (Unknown); SENS Innovation Aps (Unknown)
Responsible Party: Principal Investigator, Anna Lei Stoustrup, PhD Fellow, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPDtoParis
Record Dates: First submitted 2023-05-01; First posted 2024-02-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Telerehabilitation; COPD; Quality of Life; Mobility Limitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Mobility Limitation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Participants are anonymised with a participant identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based, longterm cycle-exercise (Experimental): One year home-based cycle exercise on a exercise bike connected to a video app from where participants can cycle push videos forward when cycling.
  Interventions: Other: Home-based cycle-exercise for COPD patients
- Standard of Care (Active Comparator): Standard of Care; exercise at fitness center, home-based exercise according to programme, self-initiated exercise
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Home-based cycle-exercise for COPD patients — Patients will cycle in their own home using a pedal exerciser connected to the 4M-video app
  Arms: Home-based, longterm cycle-exercise
Other: Standard of Care — Exercise at Fitness Center, home based exercise according to a programme
  Arms: Standard of Care

SUMMARY:
This randomised controlled trial (RCT) aims to investigate the effect of long-term, interactive home-based cycle-exercise on patients with Chronic Obstructive Pulmonary Disease (COPD) after a COPD exacerbation requiring hospitalisation. The investigators aim to investigate if patients can maintain or improve the effects of pulmonary rehabilitation in terms of walking distance, intensity of COPD symptoms, health related quality of life and Quality Adjusted Life-Years.

Participants will cycle on a pedal-exerciser in the comfort of staying in the participants' own home, whilst getting visual feedback from the 4Mvideo app. The 4Mvideo technology is a Danish designed software system, where users can cycle forward a recording of a cyclist by treading on a pedal-exerciser, thereby getting some of the experience of a real-life cycling trip at home.

The investigators will compare the clinical outcomes and daily activity levels with that of a control group consisting of COPD patients.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) have a higher risk of experiencing disability, and even though participating in pulmonary rehabilitation (PR) are efficient for regaining strength, function and relieving symptoms, effects prove difficult to maintain. Furthermore, physical attendance to outpatient PR is challenging for COPD patients, many of whom are bound to their home, due to said disability and symptoms. Even in patients who follow through with the PR programme, adherence to exercise after is a major challenge.

The investigators hypothesise that an intervention group of COPD-patients, who will receive home-based cycle exercise will maintain or even improve effects on physical fitness from PR, in terms of walking distance, daily activity levels (DAL), exercise tolerance, disease prevention and health related quality of life (HRQoL).

Furthermore, the investigators hypothesise that the participants express improved motivation in terms of adhering to exercise, when participating in home-based, interactive group cycle exercise.

It is expected to measure changes in DAL, lung function, levels of dyspnoea, exercise tolerance, walking distance, mobility, COPD symptoms, activity of daily living (ADL) related performance and HRQoL of the participants, along with assessing disease prevention. Data is compared intrapersonal and in-between groups to identify differences in outcomes at an individual level, and between intervention- and control group. Furthermore, the investigators expect to uncover identifiable in-depth insights into the values and beliefs towards exercising amongst participants.

40 participants are recruited amongst COPD patients that live in Aalborg Municipality and are admitted at Aalborg University Hospital, hospitalised due to acute exacerbation of COPD. After being discharged participants are referred to rehabilitation, for most in their own home. After rehabilitation participants are randomized into either intervention group who will exercise on exercise bikes connected with tablets in their own home. The control group will receive usual care, which consists of offers of exercising in their own home according to a programme or participating in exercise at a facility center.

ELIGIBILITY:
Inclusion Criteria:

* Adults at age > 18 years old
* Hospital admission with COPD exacerbation with pre-existing COPD diagnosis
* Citizens of Aalborg Municipality
* Able to provide informed consent
* Accepting of referral to rehabilitation

Exclusion Criteria:

* Terminal illness
* Unstable heart disease, i.e., ischemic heart disease, cardiac rhythm disorders
* Other conditions preventing participating in cycle exercise, e.g., amputation, regimens or earlier or upcoming surgeries preventing seated position, blindness
* Inability to understand basic Danish oral and written information or giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Five-repetition sit-to-stand test | Baseline measurement at initation of intervention
  The five-repetition sit-to-stand test is a test of lower limb function that measures the fastest time taken to stand five times from a chair with arms folded
Five-repetition sit-to-stand test | Changes from baseline lower limb function at follow-up are assessed at 6 weeks
  The five-repetition sit-to-stand test is a test of lower limb function that measures the fastest time taken to stand five times from a chair with arms folded
Five-repetition sit-to-stand test | Changes from baseline lower limb function at follow-up are assessed at 6 months
  The five-repetition sit-to-stand test is a test of lower limb function that measures the fastest time taken to stand five times from a chair with arms folded
Five-repetition sit-to-stand test | Changes from baseline lower limb function at follow-up are assessed at 12 months
  The five-repetition sit-to-stand test is a test of lower limb function that measures the fastest time taken to stand five times from a chair with arms folded

SECONDARY OUTCOMES:
Daily Activity Levels | Baseline measurement at initation of intervention
  Triaxial leg-mounted sensor that assesses time spent standing, walking, running, supine, cycling and sleeping/sedentary continuously throughout the day during post-hospitalisation rehabilitation for 6 weeks.
Daily Activity Levels | Changes from baseline activity during rehabilitation at follow-up are assessed 12 months
  Triaxial leg-mounted sensor that assesses time spent standing, walking, running, supine, cycling and sleeping/sedentary continuously throughout the day during post-hospitalisation rehabilitation for 6 weeks
Lung function Test (FEV1) | Baseline measurement at initation of intervention
  Forced expiratory volume in the first second in a spirometry
Lung function Test (FEV1) | Changes from baseline lung function at follow-up are assessed at 6 weeks
  Forced expiratory volume in the first second in a spirometry
Lung function Test (FEV1) | Changes from baseline lung function at follow-up are assessed at 6 months
  Forced expiratory volume in the first second in a spirometry
Lung function Test (FEV1) | Changes from baseline lung function at follow-up are assessed at 12 months
  Forced expiratory volume in the first second in a spirometry
Level of Dyspnea with the Modified Medical Research Council Dyspnoea Scale (mMRC) | Baseline measurement at initation of intervention
  A scale from 0-4 is used to assess the degree of functional disability due to dyspnoea. Higher score indicate higher degree of dyspnea
Level of Dyspnea with the Modified Medical Research Council Dyspnoea Scale (mMRC) | Changes from baseline and at follow-up are assessed at 6 weeks
  A scale from 0-4 is used to assess the degree of functional disability due to dyspnoea. Higher score indicate higher degree of dyspnea
Level of Dyspnea with the Modified Medical Research Council Dyspnoea Scale (mMRC) | Changes from baseline and at follow-up are assessed at 6 months
  A scale from 0-4 is used to assess the degree of functional disability due to dyspnoea. Higher score indicate higher degree of dyspnea
Level of Dyspnea with the Modified Medical Research Council Dyspnoea Scale (mMRC) | Changes from baseline and at follow-up are assessed at 12 months
  A scale from 0-4 is used to assess the degree of functional disability due to dyspnoea. Higher score indicate higher degree of dyspnea
Health Related Quality of Life with St. George's Respiratory Questionnaire (SGRQ) | Baseline measurement at initation of intervention
  The 2 part, 50 item questionnaire with scores from 0-100 is used to assess health impairment related to symptoms, activity, impacts, and total in patients with asthma and Chronic Obstructive Pulmonary Disease. Higher scores indicate better health related quality of life.
Health Related Quality of Life with St. George's Respiratory Questionnaire (SGRQ) | Changes from baseline health related quality of life at follow-up are assessed at 6 weeks
  The 2 part, 50 item questionnaire with scores from 0-100 is used to assess health impairment related to symptoms, activity, impacts, and total in patients with asthma and Chronic Obstructive Pulmonary Disease. Higher scores indicate better health related quality of life.
Health Related Quality of Life with St. George's Respiratory Questionnaire (SGRQ) | Changes from baseline health related quality of life at follow-up are assessed at 6 months
  The 2 part, 50 item questionnaire with scores from 0-100 is used to assess health impairment related to symptoms, activity, impacts, and total in patients with asthma and Chronic Obstructive Pulmonary Disease. Higher scores indicate better health related quality of life.
Health Related Quality of Life with St. George's Respiratory Questionnaire (SGRQ) | Changes from baseline health related quality of life at follow-up are assessed at 12 months
  The 2 part, 50 item questionnaire with scores from 0-100 is used to assess health impairment related to symptoms, activity, impacts, and total in patients with asthma and Chronic Obstructive Pulmonary Disease. Higher scores indicate better health related quality of life.
Life-Space Assessment (LSA) | Baseline measurement at initation of intervention
  Measure of performance on a range of tasks, ie. balance (score range = 0-16) and gait (score range = 0-12). Balance and gait scores are summed to produce a total score (range = 0-28) with higher scores indicate a higher degree of mobility.
Life-Space Assessment (LSA) | Changes from baseline mobility at follow-up are assessed at 6 weeks
  Measure of performance on a range of tasks, ie. balance (score range = 0-16) and gait (score range = 0-12). Balance and gait scores are summed to produce a total score (range = 0-28) with higher scores indicate a higher degree of mobility.
Life-Space Assessment (LSA) | Changes from baseline mobility at follow-up are assessed at 6 months
  Measure of performance on a range of tasks, ie. balance (score range = 0-16) and gait (score range = 0-12). Balance and gait scores are summed to produce a total score (range = 0-28) with higher scores indicate a higher degree of mobility.
Life-Space Assessment (LSA) | Changes from baseline mobility at follow-up are assessed at 12 months
  Measure of performance on a range of tasks, ie. balance (score range = 0-16) and gait (score range = 0-12). Balance and gait scores are summed to produce a total score (range = 0-28) with higher scores indicate a higher degree of mobility.
COPD Assessment Test (CAT) | Baseline measurement at initation of intervention
  Measurement of the impact of COPD on a person's life, and how this changes over time. Scale ranging from 5-30 where a higher score indicates a higher impact of COPD.
COPD Assessment Test (CAT) | Changes from baseline COPD impact at follow-up are assessed at 6 weeks
  Measurement of the impact of COPD on a person's life, and how this changes over time. Scale ranging from 5-30 where a higher score indicates a higher impact of COPD.
COPD Assessment Test (CAT) | Changes from baseline COPD impact at follow-up are assessed at 6 months
  Measurement of the impact of COPD on a person's life, and how this changes over time. Scale ranging from 5-30 where a higher score indicates a higher impact of COPD.
COPD Assessment Test (CAT) | Changes from baseline COPD impact at follow-up are assessed at 12 months
  Measurement of the impact of COPD on a person's life, and how this changes over time. Scale ranging from 5-30 where a higher score indicates a higher impact of COPD.
Tilburg Frailty Indicator (TFI) | Baseline measurement at initation of intervention
  Assessing multidimensional frailty among community-dwelling older people. Scale ranges from 0-15, with a score ranging from 0 to 8 for physical frailty, 0 to 4 for psychological frailty and 0 to 4 for social frailty. Higher scores refer to greater frailty, as older persons with a total TFI score ≥5 are considered to be frail.
Tilburg Frailty Indicator (TFI) | Changes from baseline frailty at follow-up are assessed at 6 weeks
  Assessing multidimensional frailty among community-dwelling older people. Scale ranges from 0-15, with a score ranging from 0 to 8 for physical frailty, 0 to 4 for psychological frailty and 0 to 4 for social frailty. Higher scores refer to greater frailty, as older persons with a total TFI score ≥5 are considered to be frail.
Tilburg Frailty Indicator (TFI) | Changes from baseline frailty at follow-up are assessed at 6 months
  Assessing multidimensional frailty among community-dwelling older people. Scale ranges from 0-15, with a score ranging from 0 to 8 for physical frailty, 0 to 4 for psychological frailty and 0 to 4 for social frailty. Higher scores refer to greater frailty, as older persons with a total TFI score ≥5 are considered to be frail.
Tilburg Frailty Indicator (TFI) | Changes from baseline frailty at follow-up are assessed at 12 months
  Assessing multidimensional frailty among community-dwelling older people. Scale ranges from 0-15, with a score ranging from 0 to 8 for physical frailty, 0 to 4 for psychological frailty and 0 to 4 for social frailty. Higher scores refer to greater frailty, as older persons with a total TFI score ≥5 are considered to be frail.
Clinical Frailty Scale (CFS) | Baseline measurement at initation of intervention
  Assessment of the overall level of fitness or frailty of an older adult. Scale ranges from 1-9 where a higher score indicates a higher degree of frailty.
Clinical Frailty Scale (CFS) | Changes from baseline frailty at follow-up are assessed at 6 weeks
  Assessment of the overall level of fitness or frailty of an older adult. Scale ranges from 1-9 where a higher score indicates a higher degree of frailty.
Clinical Frailty Scale (CFS) | Changes from baseline frailty at follow-up are assessed at 6 months
  Assessment of the overall level of fitness or frailty of an older adult. Scale ranges from 1-9 where a higher score indicates a higher degree of frailty.
Clinical Frailty Scale (CFS) | Changes from baseline frailty at follow-up are assessed at 12 months
  Assessment of the overall level of fitness or frailty of an older adult. Scale ranges from 1-9 where a higher score indicates a higher degree of frailty.
Canadian Occupational Performance Measure (COPM) | Baseline measurement at initation of intervention
  Qualitative outcome measure to assess a patients self-perception of performance in everyday living
Canadian Occupational Performance Measure (COPM) | Changes from baseline performance at follow-up are assessed at 6 weeks
  Qualitative outcome measure to assess a patients self-perception of performance in everyday living
Canadian Occupational Performance Measure (COPM) | Changes from baseline performance at follow-up are assessed at 6 months
  Qualitative outcome measure to assess a patients self-perception of performance in everyday living
Canadian Occupational Performance Measure (COPM) | Changes from baseline performance at follow-up are assessed at 12 months
  Qualitative outcome measure to assess a patients self-perception of performance in everyday living
Six Minutes Walk Test (6MWT) | Baseline measurement at initation of intervention
  A sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Six Minutes Walk Test (6MWT) | Changes from baseline mobility at follow-up are assessed at 6 weeks
  a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Six Minutes Walk Test (6MWT) | Changes from baseline mobility at follow-up are assessed at 6 months
  a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Six Minutes Walk Test (6MWT) | Changes from baseline and at follow-up are assessed at 12 months
  a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Short Physical Performance Battery (SPPB) | Baseline measurement at initation of intervention
  Measurement of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility.
Short Physical Performance Battery (SPPB) | Changes from baseline mobility at follow-ups are assessed at 6 weeks
  Measurement of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility.
Short Physical Performance Battery (SPPB) | Changes from baseline mobility at follow-up are assessed at 6 months
  Measurement of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility.
Short Physical Performance Battery (SPPB) | Changes from baseline mobility at follow-up are assessed at 12 months
  Measurement of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility.
Readmissions | Readmissions are assessed at 12 months
  From the electronic patient journal, data on number of participants who are readmitted, and number of individual readmissions, are collected
Survival rates | Mortality is assessed at 12 months
  From the electronic patient journal, potential deaths amongst participants are collected
EuroQol 5-Dimensions 5-Level (EQ-5D-5L) | Baseline measurement at initation of intervention
  The EQ-5D-5L test assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels ranging from "no problems" to "extreme problems." Patients select the level that best describes their health, resulting in a 5-digit number representing their health state. The EQ VAS is a separate measure where patients rate their overall health on a scale from "the best health you can imagine" to "the worst health you can imagine."
EuroQol 5-Dimensions 5-Level (EQ-5D-5L) | Changes from baseline mobility at follow-ups are assessed at 6 weeks
  The EQ-5D-5L test assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels ranging from "no problems" to "extreme problems." Patients select the level that best describes their health, resulting in a 5-digit number representing their health state. The EQ VAS is a separate measure where patients rate their overall health on a scale from "the best health you can imagine" to "the worst health you can imagine."
EuroQol 5-Dimensions 5-Level (EQ-5D-5L) | Changes from baseline mobility at follow-ups are assessed at 6 months
  The EQ-5D-5L test assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels ranging from "no problems" to "extreme problems." Patients select the level that best describes their health, resulting in a 5-digit number representing their health state. The EQ VAS is a separate measure where patients rate their overall health on a scale from "the best health you can imagine" to "the worst health you can imagine."
EuroQol 5-Dimensions 5-Level (EQ-5D-5L) | Changes from baseline mobility at follow-up are assessed at 12 months
  The EQ-5D-5L test assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels ranging from "no problems" to "extreme problems." Patients select the level that best describes their health, resulting in a 5-digit number representing their health state. The EQ VAS is a separate measure where patients rate their overall health on a scale from "the best health you can imagine" to "the worst health you can imagine."
30 Seconds Sit To Stand Test | Baseline measurement at initation of intervention
  Assessment of mobility and functional capacity, particularly in older adults or individuals with mobility impairments that measures lower body strength and endurance. The patient is asked to sit in a chair with their arms crossed over their chest and then stand up and sit down as many times as possible within 30 seconds. The total number of complete stands is recorded as the score.
30 Seconds Sit To Stand Test | Changes from baseline mobility at follow-ups are assessed at 6 weeks
  Assessment of mobility and functional capacity, particularly in older adults or individuals with mobility impairments that measures lower body strength and endurance. The patient is asked to sit in a chair with their arms crossed over their chest and then stand up and sit down as many times as possible within 30 seconds. The total number of complete stands is recorded as the score.
30 Seconds Sit To Stand Test | Changes from baseline mobility at follow-ups are assessed at 6 months
  Assessment of mobility and functional capacity, particularly in older adults or individuals with mobility impairments that measures lower body strength and endurance. The patient is asked to sit in a chair with their arms crossed over their chest and then stand up and sit down as many times as possible within 30 seconds. The total number of complete stands is recorded as the score.
30 Seconds Sit To Stand Test | Changes from baseline mobility at follow-ups are assessed at 12 months
  Assessment of mobility and functional capacity, particularly in older adults or individuals with mobility impairments that measures lower body strength and endurance. The patient is asked to sit in a chair with their arms crossed over their chest and then stand up and sit down as many times as possible within 30 seconds. The total number of complete stands is recorded as the score.

CONTACTS AND LOCATIONS:
Overall Officials: Anna L Stoustrup, MSc, Principal Investigator — a.stoustrup@rn.dk
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are accessible through enquiry to principal investigator
Supporting Information: Study Protocol
Time Frame: 01/09/2025

REFERENCES:
- [Derived] Stoustrup AL, Thomsen LP, Andreasen J, Palsson TS, Weinreich UM. Cluster randomised controlled trial on the effects of long-term home-based exercise for patients with chronic obstructive pulmonary disease with recent exacerbation: research protocol of the COPDtoParis Project. BMJ Open Respir Res. 2025 Jan 19;12(1):e002573. doi: 10.1136/bmjresp-2024-002573. PMID 39832888